CLINICAL TRIAL: NCT04629521
Title: An Observational Multicenter Clinical Study to Provide Additional Long-Term Follow-up Beyond 60 Months for Subjects Implanted With a CyPass Micro-Stent in the COMPASS Trial
Brief Title: Additional Long-Term Follow-up for Subjects Implanted With a CyPass® Micro-Stent
Acronym: COMPASS XXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GLD122-P004
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Primary Open Angle Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cataract Surgery + CyPass (Experimental): CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial)
  Interventions: Device: CyPass Micro-Stent; Procedure: Cataract Surgery

INTERVENTIONS:
Device: CyPass Micro-Stent — The CyPass Micro-Stent is a small tube with a through-lumen designed to redirect aqueous fluid from the front into the back of the eye. The device is implanted after completion of cataract surgery.
  Other Names: CyPass® Micro-Stent; Model 241-S
Procedure: Cataract Surgery — Cataract surgery involves the removal of the natural lens, which has become clouded (called a cataract), and insertion of an artificial lens (called an intraocular lens). This procedure is done through a small surgical incision in the eye.

SUMMARY:
The purpose of this study is to assess long-term (10 years post-CyPass implantation) status of the corneal endothelium in subjects who were implanted with the CyPass Micro-Stent in the COMPASS trial.

DETAILED DESCRIPTION:
The COMPASS Trial (TMI-09-01/NCT01085357) was a prospective, randomized, comparative multicenter study to assess the safety and effectiveness of the CyPass Micro-Stent in subjects with primary open angle glaucoma who were undergoing cataract surgery. In the COMPASS Trial, 374 subjects undergoing cataract surgery were randomized to the CyPass group and received the CyPass Micro-Stent, whereas 131 subjects underwent cataract surgery alone. All subjects were to be followed for 2 years postoperatively. Four hundred eighty (480) subjects completed this study.

The COMPASS XT Trial (TMI-09-01E/GLD122b-C001/NCT02700984) was designed to collect safety data beyond 24 months postoperatively for subjects who completed the COMPASS Trial. In COMPASS-XT, clinical data was collected at 36 months, 48 months, and 60 months postoperatively for a total of 5-year follow-up across the 2 studies.

In this trial, COMPASS XXT, clinical data will be collected annually for the subjects who were implanted with the CyPass Micro-Stent in the COMPASS TRIAL until the subject reaches 10 years post-CyPass implantation. For some subjects, the first visit will be at or after 10 years post-CyPass implantation, and therefore the first visit may coincide with the Exit visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Implantation with a CyPass Micro-Stent as a participant in the COMPASS trial (NCT01085357) (Transcend Medical, Incorporated, Study Number TMI-09-01).
* Able to understand the requirements of the study and willing to follow study instructions, provide written informed consent, and agree to comply with all study requirements, including the required study follow-up visits.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Inability to comply with the protocol or required follow-up visit/procedures.
* Other protocol-defined exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations Lead, Surgical, Study Director — Alcon Research, LLC
Locations (12):
- United States (12):
  - Eye Physicians and Surgeons of Arizona, Glendale, Arizona
  - Coastal Vision Medical Group, Orange, California
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Cape Coral Eye Center, Cape Coral, Florida
  - Jones Eye Center PC, Sioux City, Iowa
  - Ophthalmology Associates, St Louis, Missouri
  - Eye Associates and SurgiCenter of Vineland, Vineland, New Jersey
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Associates In Ophthalmology Ltd., West Mifflin, Pennsylvania
  - University Eye Specialists, Maryville, Tennessee
  - The Vanderbilt Eye Institute, Nashville, Tennessee
  - Ophthalmology Associates, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 12 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | Cataract Surgery + CyPass
Started | 54
Completed | 46
Not Completed | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Subject withdrew consent | 3
Not completed — Enrolled in error | 1

BASELINE CHARACTERISTICS:
Population: All enrolled
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.3 (6.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 50
  Not Reported | 1
  Unknown | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Black or African American | 6
  American Indian or Alaska Native | 0
  \Native Hawaiian or Pacific Islander | 0
  Asian | 0
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54
Endothelial Cell Density (ECD) [Mean (Standard Deviation); unit: cells per square millimeter] | 2403.93 (362.028)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Sight-threatening Adverse Events (AEs)
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (test product). This analysis was performed using data from visits in the COMPASS XXT study and includes sight-threatening adverse events as specified in the protocol. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) to Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percentage of eyes
  Persistent BCDVA loss of 3 lines or more compared to best BCDVA collected at any time during study | 18.5 [9.3 to 31.4]
  Endophthalmitis | 0.0 [0.0 to 6.6]
  Corneal decompensation | 0.0 [0.0 to 6.6]
  Retinal detachment | 0.0 [0.0 to 6.6]
  Severe choroidal hemorrhage or detachment | 0.0 [0.0 to 6.6]
  Aqueous misdirection | 0.0 [0.0 to 6.6]

2. Primary Outcome: Percentage of Eyes With Ocular Adverse Events
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (test product). This analysis was performed using data from visits in the COMPASS XXT study and includes ocular events other than sight-threatening adverse events. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) to Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percentage of eyes
  Visual Acuity Reduced | 38.9 [25.9 to 53.1]
  Visual Field Defect | 37.0 [24.3 to 51.3]
  Corneal Endothelial Cell Loss | 11.1 [4.2 to 22.6]
  Post Procedural Complication | 9.3 [3.1 to 20.3]
  Device Placement Issue | 5.6 [1.2 to 15.4]
  Hypotony Of Eye | 3.7 [0.5 to 12.7]
  Intraocular Pressure Increased | 3.7 [0.5 to 12.7]
  Optic Nerve Cup/Disc Ratio | 3.7 [0.5 to 12.7]
  Trabeculectomy | 3.7 [0.5 to 12.7]
  Cystoid Macular Oedema | 1.9 [0.0 to 9.9]
  Dermatitis | 1.9 [0.0 to 9.9]
  Device Dislocation | 1.9 [0.0 to 9.9]
  Trabeculoplasty | 1.9 [0.0 to 9.9]

3. Primary Outcome: Central Endothelial Cell Density (ECD) Reported by Mean and Standard Deviation
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. This measurement helps in monitoring the progression of corneal diseases, particularly in conditions where there is a gradual loss of endothelial cells leading to corneal edema and vision loss. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of the corneal endothelial cells in the central cornea. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed using data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: All enrolled with data at visit. Overall Number of Participants Analyzed is the number of unique subjects contributing any data to this analysis at any timepoint. In this follow-on study, not all subjects are eligible for all visits.
Measure: Mean (Standard Deviation); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
cells per millimeter squared
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 1802.49 (520.329)
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 1668.80 (707.729)
  Month 120 (Year 10): number analyzed (Participants) | 38
  Month 120 (Year 10): number analyzed (eyes) | 38
  Month 120 (Year 10) | 1574.73 (714.996)

4. Primary Outcome: Central Endothelial Cell Density (ECD) Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 3
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
cells per millimeter squared
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 1802.49 [1321.26 to 2283.71]
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 1668.80 [1448.26 to 1889.35]
  Month 120 (Year 10): number analyzed (Participants) | 38
  Month 120 (Year 10): number analyzed (eyes) | 38
  Month 120 (Year 10) | 1574.73 [1339.73 to 1809.74]

5. Primary Outcome: Central Endothelial Cell Density (ECD) Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 3
Time Frame: Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 7
Number analyzed (eyes) | 7
cells per millimeter squared
  0 percentile | 909.7
  5th percentile | 909.7
  25th percentile | 1412.5
  50th percentile | 1959.2
  75th percentile | 2185.3
  95th percentile | 2460.0
  100th percentile | 2460.0

6. Primary Outcome: Central Endothelial Cell Density (ECD) Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 3
Time Frame: Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 42
Number analyzed (eyes) | 42
cells per millimeter squared
  0 percentile | 458.8
  5th percentile | 561.0
  25th percentile | 805.7
  50th percentile | 1867.0
  75th percentile | 2222.8
  95th percentile | 2546.0
  100th percentile | 2660.8

7. Primary Outcome: Central Endothelial Cell Density (ECD) Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 3
Time Frame: Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 38
Number analyzed (eyes) | 38
cells per millimeter squared
  0 percentile | 413.5
  5th percentile | 415.7
  25th percentile | 796.6
  50th percentile | 1640.0
  75th percentile | 2165.3
  95th percentile | 2597.5
  100th percentile | 2800.8

8. Primary Outcome: Peripheral (Nasal) Endothelial Cell Density (ECD) Reported by Mean and Standard Deviation
Description: Peripheral ECD refers to the number of endothelial cells present per square millimeter in the peripheral cornea. This measurement is important for detecting peripheral corneal diseases, monitoring progression of corneal diseases, assessing the impact of contact lens wear, and ensuring optimal surgical planning (i.e., corneal transplantation). Peripheral ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of endothelial cells. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
cells per millimeter squared
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 1844.51 (684.727)
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 1739.44 (779.814)
  Month 120 (Year 10): number analyzed (Participants) | 30
  Month 120 (Year 10): number analyzed (eyes) | 30
  Month 120 (Year 10) | 1688.74 (803.605)

9. Primary Outcome: Peripheral (Nasal) Endothelial Cell Density (ECD) Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 8
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
cells per millimeter squared
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 1844.51 [1211.25 to 2477.78]
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 1739.44 [1496.44 to 1982.45]
  Month 120 (Year 10): number analyzed (Participants) | 30
  Month 120 (Year 10): number analyzed (eyes) | 30
  Month 120 (Year 10) | 1688.74 [1388.87 to 1988.61]

10. Primary Outcome: Peripheral (Nasal) Endothelial Cell Density (ECD) Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 8
Time Frame: Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 7
Number analyzed (eyes) | 7
cells per millimeter squared
  0 percentile | 489.7
  5th percentile | 489.7
  25th percentile | 1390.6
  50th percentile | 2132.7
  75th percentile | 2227.0
  95th percentile | 2465.2
  100th percentile | 2465.2

11. Primary Outcome: Peripheral (Nasal) Endothelial Cell Density (ECD) Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 8
Time Frame: Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 42
Number analyzed (eyes) | 42
cells per millimeter squared
  0 percentile | 449.5
  5th percentile | 510.0
  25th percentile | 1024.5
  50th percentile | 2020.5
  75th percentile | 2341.0
  95th percentile | 2772.0
  100th percentile | 2814.0

12. Primary Outcome: Peripheral (Nasal) Endothelial Cell Density (ECD) Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 8
Time Frame: Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 30
Number analyzed (eyes) | 30
cells per millimeter squared
  0 percentile | 353.3
  5th percentile | 477.0
  25th percentile | 856.5
  50th percentile | 1865.4
  75th percentile | 2345.5
  95th percentile | 2637.3
  100th percentile | 3183.7

13. Primary Outcome: Central Endothelial Cell Coefficient of Variation (CECCV) Reported by Mean and Standard Deviation
Description: The CECCV is a measurement used in assessing the variability and quantifying the degree of variation in endothelial cell size within the central cornea. The CECCV measurements were obtained using specular microscopy from endothelial cells within the central region of the cornea. A higher CECCV suggests greater variability in endothelial cell size within the central cornea and may suggest underlying endothelial cell pathology, such as stress, aging, or certain corneal diseases (e.g. Fuch's endothelial dystrophy). A lower CECCV indicates more uniform cell size distribution, which is typically associated with a healthier endothelial function. This analysis was performed using data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
unitless
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 28.19 (3.189)
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 29.25 (5.507)
  Month 120 (Year 10): number analyzed (Participants) | 38
  Month 120 (Year 10): number analyzed (eyes) | 38
  Month 120 (Year 10) | 30.57 (5.001)

14. Primary Outcome: Central Endothelial Cell Coefficient of Variation (CECCV) Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 13
Time Frame: Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: unitless
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 7
Number analyzed (eyes) | 7
unitless
  0 percentile | 23.8
  5th percentile | 23.8
  25th percentile | 24.8
  50th percentile | 28.2
  75th percentile | 31.0
  95th percentile | 32.3
  100th percentile | 32.3

15. Primary Outcome: Central Endothelial Cell Coefficient of Variation (CECCV) Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 13
Time Frame: Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: unitless
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 42
Number analyzed (eyes) | 42
unitless
  0 percentile | 8.0
  5th percentile | 20.5
  25th percentile | 27.0
  50th percentile | 29.4
  75th percentile | 32.2
  95th percentile | 36.3
  100th percentile | 39.5

16. Primary Outcome: Central Endothelial Cell Coefficient of Variation (CECCV) Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 13
Time Frame: Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: unitless
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 38
Number analyzed (eyes) | 38
unitless
  0 percentile | 16.5
  5th percentile | 21.5
  25th percentile | 27.8
  50th percentile | 30.8
  75th percentile | 33.8
  95th percentile | 38.8
  100th percentile | 40.5

17. Primary Outcome: Central Endothelial Hexagonality (CEH) Reported by Mean and Standard Deviation
Description: The CEH is a measurement used in assessing the regularity of endothelial cell shape within the central cornea. It provides insights into the structural integrity of the corneal endothelium, aiding in the evaluation of corneal health and diagnosis of endothelial cell-related pathologies. The CEH measurement was obtained using specular microscopy, a non-invasive imaging technique that assesses the regularity of endothelial cell shape within the central cornea. A normal cornea is of hexagonal shape. A higher CEH indicates a greater proportion of endothelial cells with a hexagonal shape, which is associated with a more regular and healthier endothelial cell morphology. A lower CEH suggests decreased hexagonality and may indicate abnormalities in endothelial cell structure or function. This analysis was performed using data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of hexagonality
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
percentage of hexagonality
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 64.33 (5.223)
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 60.96 (8.235)
  Month 120 (Year 10): number analyzed (Participants) | 38
  Month 120 (Year 10): number analyzed (eyes) | 38
  Month 120 (Year 10) | 62.09 (8.589)

18. Primary Outcome: Central Endothelial Hexagonality (CEH) Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 17
Time Frame: Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: percentage of hexagonality
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 7
Number analyzed (eyes) | 7
percentage of hexagonality
  0 percentile | 57.7
  5th percentile | 57.7
  25th percentile | 59.3
  50th percentile | 66.0
  75th percentile | 68.3
  95th percentile | 71.5
  100th percentile | 71.5

19. Primary Outcome: Central Endothelial Hexagonality (CEH) Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 17
Time Frame: Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: percentage of hexagonality
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 42
Number analyzed (eyes) | 42
percentage of hexagonality
  0 percentile | 41.0
  5th percentile | 44.3
  25th percentile | 57.8
  50th percentile | 60.8
  75th percentile | 65.7
  95th percentile | 72.5
  100th percentile | 80.7

20. Primary Outcome: Central Endothelial Hexagonality Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 17
Time Frame: Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: percentage of hexagonality
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 38
Number analyzed (eyes) | 38
percentage of hexagonality
  0 percentile | 43.3
  5th percentile | 44.0
  25th percentile | 57.8
  50th percentile | 63.4
  75th percentile | 68.2
  95th percentile | 75.8
  100th percentile | 78.3

21. Primary Outcome: Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Mean and Standard Deviation
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. This measurement helps in monitoring the progression of corneal diseases, particularly in conditions where there is a gradual loss of endothelial cells leading to corneal edema and vision loss. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of the corneal endothelial cells in the central cornea. A negative change value indicates a lessening of corneal health and function. This analysis was performed using data from the COMPASS study and data from the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
cells per millimeter squared
  Change from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Baseline at Month 96 (Year 8) | -612.31 (704.719)
  Change from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  Change from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  Change from Baseline at Month 108 (Year 9) | -762.63 (706.732)
  Change from Baseline at Month 120 (Year 10): number analyzed (Participants) | 38
  Change from Baseline at Month 120 (Year 10): number analyzed (eyes) | 38
  Change from Baseline at Month 120 (Year 10) | -819.62 (696.501)

22. Primary Outcome: Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 21
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
cells per millimeter squared
  Change from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Baseline at Month 96 (Year 8) | -612.31 [-1264.07 to 39.44]
  Change from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  Change from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  Change from Baseline at Month 108 (Year 9) | -762.63 [-982.86 to -542.39]
  Change from Baseline at Month 120 (Year 10): number analyzed (Participants) | 38
  Change from Baseline at Month 120 (Year 10): number analyzed (eyes) | 38
  Change from Baseline at Month 120 (Year 10) | -819.62 [-1048.56 to -590.69]

23. Primary Outcome: Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 21
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 7
Number analyzed (eyes) | 7
cells per millimeter squared
  0 percentile | -1802.6
  5th percentile | -1802.6
  25th percentile | -1246.7
  50th percentile | -444.5
  75th percentile | 60.2
  95th percentile | 161.8
  100th percentile | 161.8

24. Primary Outcome: Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 21
Time Frame: Baseline (COMPASS Study) preoperative, Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 42
Number analyzed (eyes) | 42
cells per millimeter squared
  0 percentile | -2028.0
  5th percentile | -1893.8
  25th percentile | -1450.1
  50th percentile | -590.3
  75th percentile | -198.3
  95th percentile | 308.0
  100th percentile | 807.6

25. Primary Outcome: Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 21
Time Frame: Baseline (COMPASS Study) preoperative, Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 38
Number analyzed (eyes) | 38
cells per millimeter squared
  0 percentile | -1937.5
  5th percentile | -1873.7
  25th percentile | -1416.4
  50th percentile | -907.6
  75th percentile | -232.0
  95th percentile | 253.8
  100th percentile | 752.1

26. Primary Outcome: Percent Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Mean and Standard Deviation
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. This measurement helps in monitoring the progression of corneal diseases, particularly in conditions where there is a gradual loss of endothelial cells leading to corneal edema and vision loss. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of the corneal endothelial cells in the central cornea. A negative percent change value indicates a worsening of corneal health and function. This analysis was performed using data from the COMPASS study and data from the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
percent change
  Change from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Baseline at Month 96 (Year 8) | -22.77 (26.468)
  Change from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  Change from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  Change from Baseline at Month 108 (Year 9) | -30.60 (31.070)
  Change from Baseline at Month 120 (Year 10): number analyzed (Participants) | 38
  Change from Baseline at Month 120 (Year 10): number analyzed (eyes) | 38
  Change from Baseline at Month 120 (Year 10) | -33.57 (31.673)

27. Primary Outcome: Percent Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 26
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent change
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
percent change
  Change from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Baseline at Month 96 (Year 8) | -22.77 [-47.25 to 1.71]
  Change from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  Change from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  Change from Baseline at Month 108 (Year 9) | -30.60 [-40.28 to -20.92]
  Change from Baseline at Month 120 (Year 10): number analyzed (Participants) | 38
  Change from Baseline at Month 120 (Year 10): number analyzed (eyes) | 38
  Change from Baseline at Month 120 (Year 10) | -33.57 [-43.98 to -23.16]

28. Primary Outcome: Percent Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 26
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: percent change
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 7
Number analyzed (eyes) | 7
percent change
  0 percentile | -66.5
  5th percentile | -66.5
  25th percentile | -46.9
  50th percentile | -16.9
  75th percentile | 3.8
  95th percentile | 7.0
  100th percentile | 7.0

29. Primary Outcome: Percent Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 26
Time Frame: Baseline (COMPASS Study) preoperative, Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: percent change
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 42
Number analyzed (eyes) | 42
percent change
  0 percentile | -79.9
  5th percentile | -74.8
  25th percentile | -65.5
  50th percentile | -24.9
  75th percentile | -8.1
  95th percentile | 18.0
  100th percentile | 50.1

30. Primary Outcome: Percent Change in Central Endothelial Cell Density (ECD) From COMPASS Trial Baseline Visit Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 26
Time Frame: Baseline (COMPASS Study) preoperative, Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: percent change
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 38
Number analyzed (eyes) | 38
percent change
  0 percentile | -81.9
  5th percentile | -80.1
  25th percentile | -61.9
  50th percentile | -35.8
  75th percentile | -8.6
  95th percentile | 16.7
  100th percentile | 46.7

31. Primary Outcome: Percentage of Eyes According to Central Endothelial Cell Density (ECD) <1000 Cells Per Millimeter Squared
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. This measurement helps in monitoring the progression of corneal diseases, particularly in conditions where there is a gradual loss of endothelial cells leading to corneal edema and vision loss. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of the corneal endothelial cells in the central cornea. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed using data from the COMPASS, COMPASS XT, and COMPASS XXT studies. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 3, Month 6, Month 12 (Year 1), Month 24 (Year 2), Month 36 (Year 3), Month 48 (Year 4), Month 60 (Year 5), Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percentage of eyes
  Month 3: number analyzed (Participants) | 52
  Month 3: number analyzed (eyes) | 52
  Month 3 | 0.0 [0.0 to 6.8]
  Month 6: number analyzed (Participants) | 53
  Month 6: number analyzed (eyes) | 53
  Month 6 | 0.0 [0.0 to 6.7]
  Month 12 (Year 1): number analyzed (Participants) | 53
  Month 12 (Year 1): number analyzed (eyes) | 53
  Month 12 (Year 1) | 0.0 [0.0 to 6.6]
  Month 24 (Year 2): number analyzed (Participants) | 53
  Month 24 (Year 2): number analyzed (eyes) | 53
  Month 24 (Year 2) | 1.9 [0.0 to 10.1]
  Month 36 (Year 3): number analyzed (Participants) | 3
  Month 36 (Year 3): number analyzed (eyes) | 3
  Month 36 (Year 3) | 0.0 [0.0 to 70.8]
  Month 48 (Year 4): number analyzed (Participants) | 31
  Month 48 (Year 4): number analyzed (eyes) | 31
  Month 48 (Year 4) | 9.7 [2.0 to 25.8]
  Month 60 (Year 5): number analyzed (Participants) | 45
  Month 60 (Year 5): number analyzed (eyes) | 45
  Month 60 (Year 5) | 6.7 [1.4 to 18.3]
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 14.3 [0.4 to 57.9]
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 26.2 [13.9 to 42.0]
  Month 120 (Year 10): number analyzed (Participants) | 38
  Month 120 (Year 10): number analyzed (eyes) | 38
  Month 120 (Year 10) | 31.6 [17.5 to 48.7]

32. Primary Outcome: Percentage of Eyes According to Central Endothelial Cell Density (ECD) <500 Cells Per Millimeter Squared
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percentage of eyes
  Month 3: number analyzed (Participants) | 52
  Month 3: number analyzed (eyes) | 52
  Month 3 | 0.0 [0.0 to 6.8]
  Month 6: number analyzed (Participants) | 53
  Month 6: number analyzed (eyes) | 53
  Month 6 | 0.0 [0.0 to 6.7]
  Month 12 (Year 1): number analyzed (Participants) | 53
  Month 12 (Year 1): number analyzed (eyes) | 53
  Month 12 (Year 1) | 0.0 [0.0 to 6.6]
  Month 24 (Year 2): number analyzed (Participants) | 53
  Month 24 (Year 2): number analyzed (eyes) | 53
  Month 24 (Year 2) | 0.0 [0.0 to 6.7]
  Month 36 (Year 3): number analyzed (Participants) | 3
  Month 36 (Year 3): number analyzed (eyes) | 3
  Month 36 (Year 3) | 0.0 [0.0 to 70.8]
  Month 48 (Year 4): number analyzed (Participants) | 31
  Month 48 (Year 4): number analyzed (eyes) | 31
  Month 48 (Year 4) | 0.0 [0.0 to 11.2]
  Month 60 (Year 5): number analyzed (Participants) | 45
  Month 60 (Year 5): number analyzed (eyes) | 45
  Month 60 (Year 5) | 0.0 [0.0 to 7.9]
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 0.0 [0.0 to 41.0]
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 2.4 [0.1 to 12.6]
  Month 120 (Year 10): number analyzed (Participants) | 38
  Month 120 (Year 10): number analyzed (eyes) | 38
  Month 120 (Year 10) | 7.9 [1.7 to 21.4]

33. Primary Outcome: Percentage of Eyes According to Central Endothelial Cell Loss (ECL) Greater Than 30 Percent From Baseline
Description: as for outcome 31
Time Frame: Baseline (COMPASS Study) preoperative, Month 3, Month 6, Month 12 (Year 1), Month 24 (Year 2), Month 36 (Year 3), Month 48 (Year 4), Month 60 (Year 5), Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percentage of eyes
  >30% Loss from Baseline at Month 3: number analyzed (Participants) | 52
  >30% Loss from Baseline at Month 3: number analyzed (eyes) | 52
  >30% Loss from Baseline at Month 3 | 9.6 [3.2 to 21.0]
  >30% Loss from Baseline at Month 6: number analyzed (Participants) | 53
  >30% Loss from Baseline at Month 6: number analyzed (eyes) | 53
  >30% Loss from Baseline at Month 6 | 9.4 [3.1 to 20.7]
  >30% Loss from Baseline at Month 12 (Year 1): number analyzed (Participants) | 53
  >30% Loss from Baseline at Month 12 (Year 1): number analyzed (eyes) | 53
  >30% Loss from Baseline at Month 12 (Year 1) | 13.0 [5.4 to 24.9]
  >30% Loss from Baseline at Month 24 (Year 2): number analyzed (Participants) | 53
  >30% Loss from Baseline at Month 24 (Year 2): number analyzed (eyes) | 53
  >30% Loss from Baseline at Month 24 (Year 2) | 9.4 [3.1 to 20.7]
  >30% Loss from Baseline at Month 36 (Year 3): number analyzed (Participants) | 3
  >30% Loss from Baseline at Month 36 (Year 3): number analyzed (eyes) | 3
  >30% Loss from Baseline at Month 36 (Year 3) | 0.0 [0.0 to 70.8]
  >30% Loss from Baseline at Month 48 (Year 4): number analyzed (Participants) | 31
  >30% Loss from Baseline at Month 48 (Year 4): number analyzed (eyes) | 31
  >30% Loss from Baseline at Month 48 (Year 4) | 19.4 [7.5 to 37.5]
  >30% Loss from Baseline at Month 60 (Year 5): number analyzed (Participants) | 45
  >30% Loss from Baseline at Month 60 (Year 5): number analyzed (eyes) | 45
  >30% Loss from Baseline at Month 60 (Year 5) | 26.7 [14.6 to 41.9]
  >30% Loss from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  >30% Loss from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  >30% Loss from Baseline at Month 96 (Year 8) | 28.6 [3.7 to 71.0]
  >30% Loss from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  >30% Loss from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  >30% Loss from Baseline at Month 108 (Year 9) | 40.5 [25.6 to 56.7]
  >30% Loss from Baseline at Month 120 (Year 10): number analyzed (Participants) | 38
  >30% Loss from Baseline at Month 120 (Year 10): number analyzed (eyes) | 38
  >30% Loss from Baseline at Month 120 (Year 10) | 52.6 [35.8 to 69.0]

34. Primary Outcome: Percentage of Eyes According to Peripheral Endothelial Cell Density (ECD) <1000 Cells Per Millimeter Squared
Description: as for outcome 8
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
percentage of eyes
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 14.3 [0.4 to 57.9]
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 23.8 [12.1 to 39.5]
  Month 120 (Year 20): number analyzed (Participants) | 30
  Month 120 (Year 20): number analyzed (eyes) | 30
  Month 120 (Year 20) | 30.0 [14.7 to 49.4]

35. Primary Outcome: Percentage of Eyes According to Peripheral Endothelial Cell Density (ECD) <500 Cells Per Millimeter Squared
Description: as for outcome 8
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 53
Number analyzed (eyes) | 53
percentage of eyes
  Month 96 (Year 8): number analyzed (Participants) | 7
  Month 96 (Year 8): number analyzed (eyes) | 7
  Month 96 (Year 8) | 14.3 [0.4 to 57.9]
  Month 108 (Year 9): number analyzed (Participants) | 42
  Month 108 (Year 9): number analyzed (eyes) | 42
  Month 108 (Year 9) | 4.8 [0.6 to 16.2]
  Month 120 (Year 20): number analyzed (Participants) | 30
  Month 120 (Year 20): number analyzed (eyes) | 30
  Month 120 (Year 20) | 6.7 [0.8 to 22.1]

36. Primary Outcome: Annualized Rate of Change in Central Endothelial Cell Density (ECD) at Each Year of Observation Reported by Mean and Standard Deviation
Description: The annualized rate of change in central ECD is used to quantify the rate at which the central ECD changes over time. The annualized rate of change in central ECD is determined by dividing the change in ECD by the duration of observation (in years). A positive annualized rate of change indicates an increase in central ECD over time, suggesting a favorable outcome or the effectiveness of interventions aimed at preserving endothelial cell density. A negative annualized rate of change signifies a decrease in central ECD, which may indicate endothelial cell loss due to factors such as aging, disease progression, or the surgical interventions. This analysis was performed using data from the COMPASS study, the COMPASS XT study, and the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Baseline (COMPASS Study) preoperative, Month 12 (Year 1), Month 24 (Year 2), Month 36 (Year 3), Month 48 (Year 4), Month 60 (Year 5), Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Mean (Standard Deviation); unit: [cells per millimeter squared] per year
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
[cells per millimeter squared] per year
  Baseline to Year 1 | -267.77 (405.731)
  Year 1 to Year 2: number analyzed (Participants) | 53
  Year 1 to Year 2: number analyzed (eyes) | 53
  Year 1 to Year 2 | -23.80 (149.533)
  Year 2 to Year 3: number analyzed (Participants) | 3
  Year 2 to Year 3: number analyzed (eyes) | 3
  Year 2 to Year 3 | -118.83 (90.832)
  Year 3 to Year 4: number analyzed (Participants) | 3
  Year 3 to Year 4: number analyzed (eyes) | 3
  Year 3 to Year 4 | -63.57 (57.630)
  Year 4 to Year 5: number analyzed (Participants) | 30
  Year 4 to Year 5: number analyzed (eyes) | 30
  Year 4 to Year 5 | -95.54 (191.951)
  Year 8 to Year 9: number analyzed (Participants) | 6
  Year 8 to Year 9: number analyzed (eyes) | 6
  Year 8 to Year 9 | -138.10 (169.597)
  Year 9 to Year 10: number analyzed (Participants) | 28
  Year 9 to Year 10: number analyzed (eyes) | 28
  Year 9 to Year 10 | -44.00 (221.290)

37. Primary Outcome: Annualized Rate of Change in Central Endothelial Cell Density (ECD) at Each Year of Observation Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 36
Time Frame: as for outcome 36
Population: All enrolled with data at visit
Measure: Mean (95% Confidence Interval); unit: [cells per millimeter squared] per year
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
[cells per millimeter squared] per year
  Baseline to Year 1 | -267.77 [-378.51 to -157.02]
  Year 1 to Year 2: number analyzed (Participants) | 53
  Year 1 to Year 2: number analyzed (eyes) | 53
  Year 1 to Year 2 | -23.80 [-65.01 to 17.42]
  Year 2 to Year 3: number analyzed (Participants) | 3
  Year 2 to Year 3: number analyzed (eyes) | 3
  Year 2 to Year 3 | -118.83 [-344.47 to 106.81]
  Year 3 to Year 4: number analyzed (Participants) | 3
  Year 3 to Year 4: number analyzed (eyes) | 3
  Year 3 to Year 4 | -63.57 [-206.73 to 79.59]
  Year 4 to Year 5: number analyzed (Participants) | 30
  Year 4 to Year 5: number analyzed (eyes) | 30
  Year 4 to Year 5 | -95.54 [-167.22 to -23.87]
  Year 8 to Year 9: number analyzed (Participants) | 6
  Year 8 to Year 9: number analyzed (eyes) | 6
  Year 8 to Year 9 | -138.10 [-316.08 to 39.88]
  Year 9 to Year 10: number analyzed (Participants) | 28
  Year 9 to Year 10: number analyzed (eyes) | 28
  Year 9 to Year 10 | -44.00 [-129.81 to 41.81]

38. Primary Outcome: Annualized Percent Rate of Change in Central Endothelial Cell Density (ECD) at Each Year of Observation Reported by Mean and Standard Deviation
Description: The annualized rate of change in central ECD is used to quantify the rate at which the central ECD changes over time. The annualized rate of change in central ECD is determined by dividing the change in ECD by the duration of observation (in years). A positive percent change per year indicates an increase in central ECD over time, suggesting a favorable outcome or the effectiveness of interventions aimed at preserving endothelial cell density. A negative percent change per year may indicate endothelial cell loss due to factors such as aging, disease progression, or the surgical interventions. This analysis was performed using data from the COMPASS study, the COMPASS XT study, and the COMPASS XXT study. Central ECD was measured in cells per millimeter squared. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: as for outcome 36
Population: All enrolled with data at visit
Measure: Mean (Standard Deviation); unit: percent change per year
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percent change per year
  Baseline to Year 1 | -10.15 (16.780)
  Year 1 to Year 2: number analyzed (Participants) | 53
  Year 1 to Year 2: number analyzed (eyes) | 53
  Year 1 to Year 2 | -1.24 (9.180)
  Year 2 to Year 3: number analyzed (Participants) | 3
  Year 2 to Year 3: number analyzed (eyes) | 3
  Year 2 to Year 3 | -4.86 (3.780)
  Year 3 to Year 4: number analyzed (Participants) | 3
  Year 3 to Year 4: number analyzed (eyes) | 3
  Year 3 to Year 4 | -2.72 (2.446)
  Year 4 to Year 5: number analyzed (Participants) | 30
  Year 4 to Year 5: number analyzed (eyes) | 30
  Year 4 to Year 5 | -5.14 (9.946)
  Year 8 to Year 9: number analyzed (Participants) | 6
  Year 8 to Year 9: number analyzed (eyes) | 6
  Year 8 to Year 9 | -8.52 (10.508)
  Year 9 to Year 10: number analyzed (Participants) | 28
  Year 9 to Year 10: number analyzed (eyes) | 28
  Year 9 to Year 10 | -2.82 (14.357)

39. Primary Outcome: Annualized Percent Rate of Change in Central Endothelial Cell Density (ECD) at Each Year of Observation Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 38
Time Frame: as for outcome 36
Population: All enrolled with data at visit
Measure: Mean (95% Confidence Interval); unit: percent change per year
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percent change per year
  Baseline to Year 1 | -10.15 [-14.73 to -5.57]
  Year 1 to Year 2: number analyzed (Participants) | 53
  Year 1 to Year 2: number analyzed (eyes) | 53
  Year 1 to Year 2 | -1.24 [-3.77 to 1.29]
  Year 2 to Year 3: number analyzed (Participants) | 3
  Year 2 to Year 3: number analyzed (eyes) | 3
  Year 2 to Year 3 | -4.86 [-14.25 to 4.53]
  Year 3 to Year 4: number analyzed (Participants) | 3
  Year 3 to Year 4: number analyzed (eyes) | 3
  Year 3 to Year 4 | -2.72 [-8.79 to 3.36]
  Year 4 to Year 5: number analyzed (Participants) | 30
  Year 4 to Year 5: number analyzed (eyes) | 30
  Year 4 to Year 5 | -5.14 [-8.85 to -1.43]
  Year 8 to Year 9: number analyzed (Participants) | 6
  Year 8 to Year 9: number analyzed (eyes) | 6
  Year 8 to Year 9 | -8.52 [-19.54 to 2.51]
  Year 9 to Year 10: number analyzed (Participants) | 28
  Year 9 to Year 10: number analyzed (eyes) | 28
  Year 9 to Year 10 | -2.82 [-8.39 to 2.74]

40. Primary Outcome: Number of Corneal Sequelae Events Associated With Endothelial Cell Loss (ECL)
Description: Corneal sequelae are occurrences of complications related to ECL in the cornea and may include corneal edema, decreased visual acuity, corneal decompensation, bullous keratopathy, etc. Corneal sequelae were quantified by counting the instances where patients experienced complications attributable to endothelial cell loss. A higher number of corneal sequelae events may indicate rapid disease progression or inadequate management of conditions leading to endothelial cell loss. A lower number of corneal sequelae events may indicate a favorable response to treatment and successful disease treatment or treatment stabilization. This analysis was performed using data from the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: corneal sequelae
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
corneal sequelae | 0

41. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Mean and Standard Deviation
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of corneal endothelial cells in the central cornea. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed using data from the COMPASS study, the COMPASS XT study, and the COMPASS XXT study. Only data for subjects with rings visible on the CyPass MicroStent device and ECD data is presented. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 3, Month 6, Month 12 (Year 1), Month 24 (Year 2), Month 36 (Year 3), Month 48 (Year 4), Month 60 (Year 5), Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells per millimeter squared
Units Other Than Participants: eyes
Groups:
- Not Visible; Lumen Only; Collar Only; 1 Ring; 2 Rings; 3 Rings: CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial)
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings | 3 Rings
Number analyzed (Participants) | 54 | 54 | 54 | 54 | 54 | 54
Number analyzed (eyes) | 54 | 54 | 54 | 54 | 54 | 54
cells per millimeter squared
  Month 3: number analyzed (Participants) | 4 | 0 | 8 | 14 | 3 | 2
  Month 3: number analyzed (eyes) | 4 | 0 | 8 | 14 | 3 | 2
  Month 3 | 1913.03 (583.158) |  | 2159.24 (467.711) | 2154.11 (309.015) | 2368.27 (306.424) | 2035.25 (7.707)
  Month 6: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  Month 6: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  Month 6 | 1769.03 (624.608) | 2394.50 (NA) — Standard deviation is undefined when there is no variability in the data | 2206.81 (383.001) | 2226.18 (324.459) | 2160.54 (309.941) | 2012.45 (66.256)
  Month 12 (Year 1): number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  Month 12 (Year 1): number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  Month 12 (Year 1) | 2000.93 (461.735) | 1756.30 (NA) — Standard deviation is undefined when there is no variability in the data | 2272.34 (345.825) | 2261.04 (394.756) | 2139.71 (307.753) | 1492.95 (293.379)
  Month 24 (Year 2): number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  Month 24 (Year 2): number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  Month 24 (Year 2) | 1938.18 (529.916) | 2449.60 (70.295) | 2189.33 (388.648) | 2144.41 (400.509) | 2186.23 (362.508) | 1309.70 (870.024)
  Month 36 (Year 3): number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 0
  Month 36 (Year 3): number analyzed (eyes) | 0 | 0 | 1 | 2 | 0 | 0
  Month 36 (Year 3) |  |  | 2324.50 (NA) — Standard deviation is undefined when there is no variability in the data | 2338.00 (199.121) |  |
  Month 48 (Year 4): number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  Month 48 (Year 4): number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  Month 48 (Year 4) | 2062.20 (364.440) | 2555.70 (NA) — Standard deviation is undefined when there is no variability in the data | 2307.67 (280.270) | 2117.21 (301.552) | 1616.86 (601.855) | 742.00 (36.062)
  Month 60 (Year 5): number analyzed (Participants) | 6 | 2 | 12 | 13 | 10 | 0
  Month 60 (Year 5): number analyzed (eyes) | 6 | 2 | 12 | 13 | 10 | 0
  Month 60 (Year 5) | 2292.05 (381.087) | 2342.00 (27.577) | 2159.78 (375.998) | 2016.68 (495.751) | 1645.16 (433.827) |
  Month 96 (Year 8): number analyzed (Participants) | 1 | 1 | 1 | 2 | 2 | 0
  Month 96 (Year 8): number analyzed (eyes) | 1 | 1 | 1 | 2 | 2 | 0
  Month 96 (Year 8) | 1660.70 (NA) — Standard deviation is undefined when there is no variability in the data | 1412.50 (NA) — Standard deviation is undefined when there is no variability in the data | 2185.30 (NA) — Standard deviation is undefined when there is no variability in the data | 2209.60 (354.119) | 1469.85 (792.172) |
  Month 108 (Year 9): number analyzed (Participants) | 9 | 4 | 10 | 11 | 6 | 0
  Month 108 (Year 9): number analyzed (eyes) | 9 | 4 | 10 | 11 | 6 | 0
  Month 108 (Year 9) | 1894.88 (639.384) | 1735.63 (232.046) | 2049.77 (585.452) | 1720.05 (740.783) | 925.40 (401.250) |
  Month 120 (Year 10): number analyzed (Participants) | 6 | 7 | 9 | 9 | 5 | 0
  Month 120 (Year 10): number analyzed (eyes) | 6 | 7 | 9 | 9 | 5 | 0
  Month 120 (Year 10) | 1897.05 (730.546) | 1663.71 (593.233) | 1941.97 (661.397) | 1486.70 (721.315) | 924.90 (421.601) |

42. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 3
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of corneal endothelial cells in the central cornea. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed using data from the COMPASS study. Only data for subjects with rings visible on the CyPass MicroStent device and ECD data is presented. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 3 postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Collar Only | 1 Ring | 2 Rings | 3 Rings
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31
Number analyzed (eyes) | 31 | 31 | 31 | 31 | 31
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  0 percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  0 percentile | 1364.2 | 1230.3 | 1592.5 | 2179.0 | 2029.8
  5th percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  5th percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  5th percentile | 1364.2 | 1230.3 | 1592.5 | 2179.0 | 2029.8
  25th percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  25th percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  25th percentile | 1409.5 | 1879.4 | 2025.1 | 2179.0 | 2029.8
  50th percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  50th percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  50th percentile | 1920.0 | 2361.3 | 2171.5 | 2204.0 | 2035.3
  75th percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  75th percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  75th percentile | 2416.6 | 2506.3 | 2351.5 | 2721.8 | 2040.7
  95th percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  95th percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  95th percentile | 2447.9 | 2549.8 | 2600.8 | 2721.8 | 2040.7
  100th percentile: number analyzed (Participants) | 4 | 8 | 14 | 3 | 2
  100th percentile: number analyzed (eyes) | 4 | 8 | 14 | 3 | 2
  100th percentile | 2447.9 | 2549.8 | 2600.8 | 2721.8 | 2040.7

43. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 6
Description: as for outcome 42
Time Frame: Month 6 postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings | 3 Rings
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 34
Number analyzed (eyes) | 34 | 34 | 34 | 34 | 34 | 34
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  0 percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  0 percentile | 1361.1 | 2394.5 | 1418.0 | 1672.0 | 1693.7 | 1965.6
  5th percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  5th percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  5th percentile | 1361.1 | 2394.5 | 1418.0 | 1672.0 | 1693.7 | 1965.6
  25th percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  25th percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  25th percentile | 1361.1 | 2394.5 | 2043.0 | 2109.2 | 1899.7 | 1965.6
  50th percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  50th percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  50th percentile | 1457.9 | 2394.5 | 2337.7 | 2257.5 | 2248.6 | 2012.5
  75th percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  75th percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  75th percentile | 2488.1 | 2394.5 | 2463.9 | 2558.3 | 2304.3 | 2059.3
  95th percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  95th percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  95th percentile | 2488.1 | 2394.5 | 2547.5 | 2662.3 | 2650.8 | 2059.3
  100th percentile: number analyzed (Participants) | 3 | 1 | 8 | 13 | 7 | 2
  100th percentile: number analyzed (eyes) | 3 | 1 | 8 | 13 | 7 | 2
  100th percentile | 2488.1 | 2394.5 | 2547.5 | 2662.3 | 2650.8 | 2059.3

44. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 12 (Year 1)
Description: as for outcome 42
Time Frame: Month 12 (Year 1) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings | 3 Rings
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48 | 48
Number analyzed (eyes) | 48 | 48 | 48 | 48 | 48 | 48
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  0 percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  0 percentile | 1357.7 | 1756.3 | 1388.7 | 1340.5 | 1659.6 | 1285.5
  5th percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  5th percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  5th percentile | 1357.7 | 1756.3 | 1388.7 | 1531.0 | 1659.6 | 1285.5
  25th percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  25th percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  25th percentile | 1666.8 | 1756.3 | 2146.8 | 2125.7 | 1907.0 | 1285.5
  50th percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  50th percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  50th percentile | 2139.9 | 1756.3 | 2414.8 | 2359.3 | 2234.2 | 1493.0
  75th percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  75th percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  75th percentile | 2335.1 | 1756.3 | 2480.7 | 2563.3 | 2293.8 | 1700.4
  95th percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  95th percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  95th percentile | 2366.3 | 1756.3 | 2579.2 | 2666.0 | 2588.2 | 1700.4
  100th percentile: number analyzed (Participants) | 4 | 1 | 12 | 21 | 8 | 2
  100th percentile: number analyzed (eyes) | 4 | 1 | 12 | 21 | 8 | 2
  100th percentile | 2366.3 | 1756.3 | 2579.2 | 2852.3 | 2588.2 | 1700.4

45. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 24 (Year 2)
Description: as for outcome 42
Time Frame: Month 24 (Year 2) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings | 3 Rings
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50 | 50
Number analyzed (eyes) | 50 | 50 | 50 | 50 | 50 | 50
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  0 percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  0 percentile | 1350.2 | 2370.2 | 1301.3 | 1526.7 | 1390.0 | 694.5
  5th percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  5th percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  5th percentile | 1350.2 | 2370.2 | 1301.3 | 1526.7 | 1390.0 | 694.5
  25th percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  25th percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  25th percentile | 1432.2 | 2370.2 | 1961.0 | 1721.2 | 2071.9 | 694.5
  50th percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  50th percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  50th percentile | 2047.7 | 2474.7 | 2345.9 | 2152.7 | 2226.4 | 1309.7
  75th percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  75th percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  75th percentile | 2318.7 | 2503.9 | 2443.3 | 2503.2 | 2373.1 | 1924.9
  95th percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  95th percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  95th percentile | 2542.1 | 2503.9 | 2624.5 | 2757.6 | 2732.7 | 1924.9
  100th percentile: number analyzed (Participants) | 5 | 3 | 12 | 16 | 12 | 2
  100th percentile: number analyzed (eyes) | 5 | 3 | 12 | 16 | 12 | 2
  100th percentile | 2542.1 | 2503.9 | 2624.5 | 2757.6 | 2732.7 | 1924.9

46. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 36 (Year 3)
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of corneal endothelial cells in the central cornea. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed using data from the COMPASS XT study. Only data for subjects with rings visible on the CyPass MicroStent device and ECD data is presented. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 36 (Year 3) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Collar Only | 1 Ring
Number analyzed (Participants) | 3 | 3
Number analyzed (eyes) | 3 | 3
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 1 | 2
  0 percentile: number analyzed (eyes) | 1 | 2
  0 percentile | 2324.5 | 2197.2
  5th percentile: number analyzed (Participants) | 1 | 2
  5th percentile: number analyzed (eyes) | 1 | 2
  5th percentile | 2324.5 | 2197.2
  25th percentile: number analyzed (Participants) | 1 | 2
  25th percentile: number analyzed (eyes) | 1 | 2
  25th percentile | 2324.5 | 2197.2
  50th percentile: number analyzed (Participants) | 1 | 2
  50th percentile: number analyzed (eyes) | 1 | 2
  50th percentile | 2324.5 | 2338.0
  75th percentile: number analyzed (Participants) | 1 | 2
  75th percentile: number analyzed (eyes) | 1 | 2
  75th percentile | 2324.5 | 2478.8
  95th percentile: number analyzed (Participants) | 1 | 2
  95th percentile: number analyzed (eyes) | 1 | 2
  95th percentile | 2324.5 | 2478.8
  100th percentile: number analyzed (Participants) | 1 | 2
  100th percentile: number analyzed (eyes) | 1 | 2
  100th percentile | 2324.5 | 2478.8

47. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 48 (Year 4)
Description: as for outcome 46
Time Frame: Month 48 (Year 4) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings | 3 Rings
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31
Number analyzed (eyes) | 31 | 31 | 31 | 31 | 31 | 31
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  0 percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  0 percentile | 1684.7 | 2555.7 | 1678.7 | 1524.0 | 752.5 | 716.5
  5th percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  5th percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  5th percentile | 1684.7 | 2555.7 | 1678.7 | 1524.0 | 752.5 | 716.5
  25th percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  25th percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  25th percentile | 1684.7 | 2555.7 | 2304.0 | 2034.8 | 1468.8 | 716.5
  50th percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  50th percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  50th percentile | 2089.9 | 2555.7 | 2334.0 | 2107.5 | 1550.2 | 742.0
  75th percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  75th percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  75th percentile | 2412.0 | 2555.7 | 2475.2 | 2375.3 | 1940.5 | 767.5
  95th percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  95th percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  95th percentile | 2412.0 | 2555.7 | 2683.7 | 2537.5 | 2372.3 | 767.5
  100th percentile: number analyzed (Participants) | 3 | 1 | 9 | 11 | 5 | 2
  100th percentile: number analyzed (eyes) | 3 | 1 | 9 | 11 | 5 | 2
  100th percentile | 2412.0 | 2555.7 | 2683.7 | 2537.5 | 2372.3 | 767.5

48. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 60 (Year 5)
Description: as for outcome 46
Time Frame: Month 60 (Year 5) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 43 | 43 | 43 | 43 | 43
Number analyzed (eyes) | 43 | 43 | 43 | 43 | 43
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  0 percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  0 percentile | 1683.7 | 2322.5 | 1345.3 | 1109.0 | 741.7
  5th percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  5th percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  5th percentile | 1683.7 | 2322.5 | 1345.3 | 1109.0 | 741.7
  25th percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  25th percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  25th percentile | 2050.2 | 2322.5 | 2080.0 | 1734.2 | 1372.0
  50th percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  50th percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  50th percentile | 2342.7 | 2342.0 | 2277.9 | 2035.8 | 1743.6
  75th percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  75th percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  75th percentile | 2589.3 | 2361.5 | 2411.7 | 2417.7 | 1912.5
  95th percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  95th percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  95th percentile | 2743.8 | 2361.5 | 2555.8 | 2958.7 | 2242.5
  100th percentile: number analyzed (Participants) | 6 | 2 | 12 | 13 | 10
  100th percentile: number analyzed (eyes) | 6 | 2 | 12 | 13 | 10
  100th percentile | 2743.8 | 2361.5 | 2555.8 | 2958.7 | 2242.5

49. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 96 (Year 8)
Description: Central ECD refers to the number of endothelial cells present per square millimeter in the central cornea. Central ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of corneal endothelial cells in the central cornea. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed using data from the COMPASS XXT study. Only data for subjects with rings visible on the CyPass MicroStent device and ECD data is presented. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
Number analyzed (eyes) | 7 | 7 | 7 | 7 | 7
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  0 percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  0 percentile | 1660.7 | 1412.5 | 2185.3 | 1959.2 | 909.7
  5th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  5th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  5th percentile | 1660.7 | 1412.5 | 2185.3 | 1959.2 | 909.7
  25th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  25th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  25th percentile | 1660.7 | 1412.5 | 2185.3 | 1959.2 | 909.7
  50th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  50th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  50th percentile | 1660.7 | 1412.5 | 2185.3 | 2209.6 | 1469.9
  75th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  75th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  75th percentile | 1660.7 | 1412.5 | 2185.3 | 2460.0 | 2030.0
  95th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  95th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  95th percentile | 1660.7 | 1412.5 | 2185.3 | 2460.0 | 2030.0
  100th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  100th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  100th percentile | 1660.7 | 1412.5 | 2185.3 | 2460.0 | 2030.0

50. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 49
Time Frame: Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40
Number analyzed (eyes) | 40 | 40 | 40 | 40 | 40
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  0 percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  0 percentile | 547.5 | 1438.5 | 699.3 | 458.8 | 568.3
  5th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  5th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  5th percentile | 547.5 | 1438.5 | 699.3 | 458.8 | 568.3
  25th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  25th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  25th percentile | 1612.0 | 1583.6 | 2131.3 | 805.7 | 684.3
  50th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  50th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  50th percentile | 2180.7 | 1750.1 | 2217.2 | 2014.7 | 783.7
  75th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  75th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  75th percentile | 2222.8 | 1887.7 | 2362.5 | 2301.0 | 1057.7
  95th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  95th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  95th percentile | 2573.2 | 2003.8 | 2660.8 | 2546.0 | 1674.8
  100th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  100th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  100th percentile | 2573.2 | 2003.8 | 2660.8 | 2546.0 | 1674.8

51. Primary Outcome: Central Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 49
Time Frame: Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36
Number analyzed (eyes) | 36 | 36 | 36 | 36 | 36
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  0 percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  0 percentile | 483.5 | 796.6 | 624.7 | 413.5 | 415.7
  5th percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  5th percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  5th percentile | 483.5 | 796.6 | 624.7 | 413.5 | 415.7
  25th percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  25th percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  25th percentile | 1881.9 | 951.7 | 1503.2 | 782.7 | 640.3
  50th percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  50th percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  50th percentile | 2121.0 | 1849.5 | 2165.3 | 1637.8 | 966.0
  75th percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  75th percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  75th percentile | 2177.4 | 2102.7 | 2359.1 | 1960.5 | 1094.2
  95th percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  95th percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  95th percentile | 2597.5 | 2363.3 | 2800.8 | 2479.7 | 1508.3
  100th percentile: number analyzed (Participants) | 6 | 7 | 9 | 9 | 5
  100th percentile: number analyzed (eyes) | 6 | 7 | 9 | 9 | 5
  100th percentile | 2597.5 | 2363.3 | 2800.8 | 2479.7 | 1508.3

52. Primary Outcome: Peripheral Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Mean and Standard Deviation
Description: Peripheral ECD refers to the number of endothelial cells present per square millimeter in the peripheral cornea. Peripheral ECD was assessed using specular microscopy, a non-invasive imaging technique that allows for visualization and quantification of endothelial cells. A normal ECD in adults typically ranges between 2500 to 3000 cells per square millimeter, although this can vary depending on age and individual variation. A higher value indicates better corneal health and function. A lower value suggests potential endothelial dysfunction or damage. This analysis was performed data from visits in the COMPASS XXT study. Only data for subjects with rings visible on the CyPass MicroStent device and ECD data is presented. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48
Number analyzed (eyes) | 48 | 48 | 48 | 48 | 48
cells per millimeter squared
  Month 96 (Year 8): number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  Month 96 (Year 8): number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  Month 96 (Year 8) | 2132.70 (NA) — Standard deviation is undefined when there is no variability in the data | 1390.60 (NA) — Standard deviation is undefined when there is no variability in the data | 2227.00 (NA) — Standard deviation is undefined when there is no variability in the data | 2103.20 (152.028) | 1477.45 (1396.889)
  Month 108 (Year 9): number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  Month 108 (Year 9): number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  Month 108 (Year 9) | 2062.49 (728.658) | 1828.05 (399.061) | 2087.86 (599.144) | 1752.28 (835.401) | 915.63 (585.915)
  Month 120 (Year 10): number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  Month 120 (Year 10): number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  Month 120 (Year 10) | 2177.90 (988.439) | 1955.98 (348.144) | 1663.57 (730.987) | 1683.19 (909.922) | 976.46 (550.677)

53. Primary Outcome: Peripheral Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 96 (Year 8)
Description: as for outcome 52
Time Frame: Month 96 (Year 8) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
Number analyzed (eyes) | 7 | 7 | 7 | 7 | 7
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  0 percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  0 percentile | 2132.7 | 1390.6 | 2227.0 | 1995.7 | 489.7
  5th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  5th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  5th percentile | 2132.7 | 1390.6 | 2227.0 | 1995.7 | 489.7
  25th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  25th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  25th percentile | 2132.7 | 1390.6 | 2227.0 | 1995.7 | 489.7
  50th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  50th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  50th percentile | 2132.7 | 1390.6 | 2227.0 | 2103.2 | 1477.5
  75th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  75th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  75th percentile | 2132.7 | 1390.6 | 2227.0 | 2210.7 | 2465.2
  95th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  95th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  95th percentile | 2132.7 | 1390.6 | 2227.0 | 2210.7 | 2465.2
  100th percentile: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
  100th percentile: number analyzed (eyes) | 1 | 1 | 1 | 2 | 2
  100th percentile | 2132.7 | 1390.6 | 2227.0 | 2210.7 | 2465.2

54. Primary Outcome: Peripheral Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 108 (Year 9)
Description: as for outcome 52
Time Frame: Month 108 (Year 9) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40
Number analyzed (eyes) | 40 | 40 | 40 | 40 | 40
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  0 percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  0 percentile | 516.5 | 1373.0 | 569.0 | 449.5 | 479.2
  5th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  5th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  5th percentile | 516.5 | 1373.0 | 569.0 | 449.5 | 479.2
  25th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  25th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  25th percentile | 1848.4 | 1575.9 | 2106.0 | 803.8 | 514.8
  50th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  50th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  50th percentile | 2272.0 | 1796.7 | 2262.3 | 2037.3 | 633.6
  75th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  75th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  75th percentile | 2515.5 | 2080.3 | 2331.2 | 2483.8 | 1283.2
  95th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  95th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  95th percentile | 2814.0 | 2345.8 | 2784.7 | 2772.0 | 1949.5
  100th percentile: number analyzed (Participants) | 9 | 4 | 10 | 11 | 6
  100th percentile: number analyzed (eyes) | 9 | 4 | 10 | 11 | 6
  100th percentile | 2814.0 | 2345.8 | 2784.7 | 2772.0 | 1949.5

55. Primary Outcome: Peripheral Endothelial Cell Density (ECD) by Number of Rings Observed at the Visit Reported by Percentile - Month 120 (Year 10)
Description: as for outcome 52
Time Frame: Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: cells per millimeter squared
Units Other Than Participants: eyes
Arm/Group | Not Visible | Lumen Only | Collar Only | 1 Ring | 2 Rings
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
Number analyzed (eyes) | 30 | 30 | 30 | 30 | 30
cells per millimeter squared
  0 percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  0 percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  0 percentile | 526.5 | 1512.7 | 647.7 | 477.0 | 353.3
  5th percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  5th percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  5th percentile | 526.5 | 1512.7 | 647.7 | 477.0 | 353.3
  25th percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  25th percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  25th percentile | 2262.8 | 1695.8 | 922.5 | 683.0 | 643.2
  50th percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  50th percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  50th percentile | 2408.8 | 2042.5 | 1709.8 | 2080.0 | 856.5
  75th percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  75th percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  75th percentile | 2507.7 | 2157.6 | 2250.2 | 2412.6 | 1269.8
  95th percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  95th percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  95th percentile | 3183.7 | 2371.3 | 2597.0 | 2637.3 | 1759.5
  100th percentile: number analyzed (Participants) | 5 | 5 | 7 | 8 | 5
  100th percentile: number analyzed (eyes) | 5 | 5 | 7 | 8 | 5
  100th percentile | 3183.7 | 2371.3 | 2597.0 | 2637.3 | 1759.5

56. Primary Outcome: Number of Secondary Surgical Intervention (SSI) Events to Modify the Device Position (eg, Repositioning, Trimming, Explantation)
Description: SSI events are additional surgical procedures performed after the initial placement of the CyPass micro-stent device to adjust its position or address issues related to its placement. SSI were noted through adverse event reporting, clinical evaluation, comprehensive documentation of outcome assessment and data analysis. A higher number of SSI events may indicate challenges or complications related to the initial placement of the CyPass device, technical difficulties during the initial surgery, device-related issues, or patient-specific factors contributing to the need for additional interventions. A lower number of SSI events may suggest that the initial device placement was successful and well-tolerated, with fewer complications or the need for adjustments. This analysis was performed using data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) to Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: secondary surgical interventions
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
secondary surgical interventions | 0

57. Primary Outcome: Percentage of Eyes With CyPass Micro-Stent Movement and/or Malposition
Description: CyPass micro-stent movement and/or malposition refers to issues related to the displacement or improper positioning of the CyPass Micro-Stent in the eye's drainage angle. The investigator qualitatively and subjectively assessed the position of the device by counting the visible number of rings of the device during a gonioscopic exam, which used a specialized lens to visually assess the position and stability of the CyPass device. Movement and/or malposition may suggest a greater risk of complications or inadequate treatment of glaucoma. This analysis was performed using data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) to Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
percentage of eyes | 7.4 [2.1 to 17.9]

58. Primary Outcome: Number of Corneal Adverse Events Caused by CyPass MicroStent
Description: A corneal adverse event is an undesirable occurrence related to the cornea, such as inflammation, edema, epithelial defects, or other complications. The number of corneal adverse events caused by the CyPass Micro-Stent was assessed from patient reporting, clinical observation and documentation during patients' follow-up visits. This analysis was performed using data from visits in the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) to Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: events
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
events | 0

59. Primary Outcome: Number of Events of Best Corrected Visual Acuity (BCVA) Loss of 10 Letters or More
Description: Visual acuity was measured with correction in place using letter charts. BCVA [synonymous with Best Corrected Distance Visual Acuity (BCDVA)] at each visit was compared to the participant's best achieved BCVA recorded throughout the 10-year period after CyPass implantation. This analysis was performed using data from the COMPASS study, the COMPASS XT study, and the COMPASS XXT study. No hypothesis testing was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Month 96 (Year 8) to Month 120 (Year 10) postoperative
Population: All enrolled with data at visit
Measure: Number; unit: events
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
events | 21

60. Primary Outcome: Change in Visual Field Mean Deviation From COMPASS Trial Screening Visit Reported by Mean and Standard Deviation
Description: Visual field mean deviation is a measure used in visual field testing to assess the overall sensitivity of a patient's vision compared to a standardized norm. The Humphrey automated perimeter with the 24-2 Swedish Interactive Thresholding Algorithm (SITA) standard testing method was used. Deviations were recorded in decibels. Normal deviation values are typically within 0 to -2 decibels (dB). A more negative number indicates decreased sensitivity and worsening of the overall visual field. This analysis was performed using data from the COMPASS study and data from the COMPASS XXT study. No hypothesis was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Screening (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: decibel
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
decibel
  Change from Screening Visit at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Screening Visit at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Screening Visit at Month 96 (Year 8) | 2.379 (3.7404)
  Change from Screening Visit at Month 108 (Year 9): number analyzed (Participants) | 41
  Change from Screening Visit at Month 108 (Year 9): number analyzed (eyes) | 41
  Change from Screening Visit at Month 108 (Year 9) | -1.176 (6.1884)
  Change from Screening Visit at Month 120 (Year 10): number analyzed (Participants) | 46
  Change from Screening Visit at Month 120 (Year 10): number analyzed (eyes) | 46
  Change from Screening Visit at Month 120 (Year 10) | -2.321 (4.6707)

61. Primary Outcome: Percentage of Eyes With Change in Visual Field Mean Deviation From COMPASS Trial Screening Visit Reported Categorically - 2 Decibel (dB)
Description: Visual field mean deviation is a measure used in visual field testing to assess the overall sensitivity of a patient's vision compared to a standardized norm. The Humphrey automated perimeter with the 24-2 SITA standard testing method was used. Deviations were recorded in decibels. Normal deviation values are typically within 0 to -2 decibels (dB). A more negative number indicates decreased sensitivity and worsening of the overall visual field. This analysis was performed using data from the COMPASS study and data from the COMPASS XXT study. No hypothesis was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Screening (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Increase > 2.0 dB; No Change (-2.0 dB to 2.0 dB); Decrease > 2.0 dB: CyPass Micro-Stent implanted at the conclusion of cataract surgery (COMPASS trial)
Arm/Group | Increase > 2.0 dB | No Change (-2.0 dB to 2.0 dB) | Decrease > 2.0 dB
Number analyzed (Participants) | 54 | 54 | 54
Number analyzed (eyes) | 54 | 54 | 54
percentage of eyes
  Change from Screening Visit at Month 96 (Year 8): number analyzed (Participants) | 7 | 7 | 7
  Change from Screening Visit at Month 96 (Year 8): number analyzed (eyes) | 7 | 7 | 7
  Change from Screening Visit at Month 96 (Year 8) | 42.9 | 51.7 | 0.0
  Change from Screening Visit at Month 108 (Year 9): number analyzed (Participants) | 41 | 41 | 41
  Change from Screening Visit at Month 108 (Year 9): number analyzed (eyes) | 41 | 41 | 41
  Change from Screening Visit at Month 108 (Year 9) | 9.8 | 51.2 | 39.0
  Change from Screening Visit at Month 120 (Year 10): number analyzed (Participants) | 46 | 46 | 46
  Change from Screening Visit at Month 120 (Year 10): number analyzed (eyes) | 46 | 46 | 46
  Change from Screening Visit at Month 120 (Year 10) | 10.9 | 45.7 | 43.5

62. Primary Outcome: Change in Central Corneal Thickness (CCT) From COMPASS Trial Baseline Visit Reported by Mean and Standard Deviation
Description: CCT is a measurement of the thickness of the cornea at its center and is assessed using a procedure called corneal pachymetry. A high CCT (thick cornea) indicates a central cornea thicker than average and may be associated with conditions such as corneal edema, Fuchs' dystrophy, or ocular hypertension. A low CCT (thin cornea) indicates a central cornea thinner than average and may be a risk factor for developing conditions such as glaucoma. A negative change value indicates a decrease in corneal thickness. This analysis was performed using data from the COMPASS study and data from the COMPASS XXT study. No hypothesis was prespecified for this outcome measure. One eye (study eye) contributed data to this analysis.
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
microns
  Change from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Baseline at Month 96 (Year 8) | 1.9 (22.08)
  Change from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  Change from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  Change from Baseline at Month 108 (Year 9) | 0.0 (22.84)
  Change from Baseline at Month 120 (Year 10): number analyzed (Participants) | 46
  Change from Baseline at Month 120 (Year 10): number analyzed (eyes) | 46
  Change from Baseline at Month 120 (Year 10) | 4.1 (25.09)

63. Primary Outcome: Change in Central Corneal Thickness (CCT) From COMPASS Trial Baseline Visit Reported by Mean and 95 Percent Confidence Interval
Description: as for outcome 62
Time Frame: Baseline (COMPASS Study) preoperative, Month 96 (Year 8), Month 108 (Year 9), Month 120 (Year 10) postoperative
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: microns
Units Other Than Participants: eyes
Arm/Group | Cataract Surgery + CyPass
Number analyzed (Participants) | 54
Number analyzed (eyes) | 54
microns
  Change from Baseline at Month 96 (Year 8): number analyzed (Participants) | 7
  Change from Baseline at Month 96 (Year 8): number analyzed (eyes) | 7
  Change from Baseline at Month 96 (Year 8) | 1.9 [-18.6 to 22.3]
  Change from Baseline at Month 108 (Year 9): number analyzed (Participants) | 42
  Change from Baseline at Month 108 (Year 9): number analyzed (eyes) | 42
  Change from Baseline at Month 108 (Year 9) | 0.0 [-7.1 to 7.1]
  Change from Baseline at Month 120 (Year 10): number analyzed (Participants) | 46
  Change from Baseline at Month 120 (Year 10): number analyzed (eyes) | 46
  Change from Baseline at Month 120 (Year 10) | 4.1 [-3.4 to 11.5]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent (COMPASS XXT) until time of study exit (COMPASS XXT), from 1 day to 2 years depending on point of enrollment.
Description: This analysis population includes all enrolled subjects. Safety was assessed at each visit. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more arms.
Groups:
- Cataract Surgery + CyPass - Ocular Adverse Events: Adverse events reported in this group occurred in the study eye
- Cataract Surgery + CyPass - Systemic Adverse Events: Adverse events reported in this group occurred systemically and include adverse events in the non-study eye
Arm/Group | Cataract Surgery + CyPass - Ocular Adverse Events | Cataract Surgery + CyPass - Systemic Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/54 | 1/54
Serious Adverse Events (participants affected / at risk) | 12/54 | 2/54
Other Adverse Events (participants affected / at risk) | 31/54 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cataract Surgery + CyPass - Ocular Adverse Events (N=54) | Cataract Surgery + CyPass - Systemic Adverse Events (N=54)
Visual Acuity Reduced (Eye disorders) | 10 (10) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Visual Field Defect (Nervous system disorders) | 2 (2) | 0 (0)
Trabeculectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Trabeculoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) — Non-study eye
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cataract Surgery + CyPass - Ocular Adverse Events (N=54) | Cataract Surgery + CyPass - Systemic Adverse Events (N=54)
Corneal Endothelial Cell Loss (Eye disorders) | 6 (6) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 14 (14) | 0 (0)
Device Placement Issue (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Visual Field Defect (Nervous system disorders) | 18 (18) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04629521/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04629521/SAP_001.pdf